CLINICAL TRIAL: NCT04889313
Title: Neurologic Symptoms After Non-severe COVID-19 : Analysis and Diagnosis Assessment of Somatic Spectrum Disorder
Brief Title: Post COVID-19 Neurologic Symptoms : a Somatic Spectrum Disorder ? (SOMATiC)
Acronym: SOMATiC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_NEURO_01
Record Dates: First submitted 2021-05-14; First posted 2021-05-17 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: Somatic Symptom Disorder; COVID-19; Neurologic symptoms
MeSH Terms: conditions — COVID-19; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A growing number of studies highlight the persistence of symptoms after the acute phase of SARS-CoV-2 infection, including in outpatients with mild to moderate forms of the disease. More than 80% of patients with persistent post-COVID-19 symptoms reported neurologic and neurocognitive disturbances. The pathophysiological mechanism is currently unknown, and several hypotheses have been put forward. Involvement of a Somatic Symptom Disorder (SSD) is plausible given the similarity of these symptoms with the Chronic Fatigue Syndrome identified as a SSD subtype. The objective of the SOMATiC study (SOMAtic symptom disorders Triggered by COVID-19) is to determine whether a positive diagnosis of SSD can be asserted in patients with persistent post-COVID-19 neurological symptoms.

DETAILED DESCRIPTION:
A growing number of studies highlight the persistence of symptoms after the acute phase of SARS-CoV-2 infection, including in outpatients with mild to moderate forms of the disease. More than 80% of patients with persistent post-COVID-19 symptoms reported neurologic and neurocognitive disturbances. The pathophysiological mechanism is currently unknown, and several hypotheses have been put forward. Involvement of a Somatic Symptom Disorder (SSD) is plausible given the similarity of these symptoms with the Chronic Fatigue Syndrome identified as a SSD subtype. The objective of the SOMATiC study (SOMAtic symptom disorders Triggered by COVID-19) is to determine whether a positive diagnosis of SSD can be asserted in patients with persistent post-COVID-19 neurological symptoms. The study includes consecutive patients referred for neurology consultation because of chronic neurologic symptoms after the acute phase of COVID-19. Data are collected with medical record and by phone interview. It consisted of a semi-structured interview followed by hetero-assessed scales. A positive diagnosis of SSD was established with all the following criteria: a PHQ15 score greater than or equal to 12 (criterion A); an SSD12 score greater than or equal to 23 (criterion B); an evolution of symptoms greater than or equal to four weeks for criterion C. To complete the DSMV criteria, the investigators assessed the presence of indirect argument in favor of SSD diagnosis : a traumatic experience of the initial episode collected during the interview, post-traumatic stress disorder measured by the IES-R scale, a psychiatric history collected during the interview, significant alexithymia measured by the TAS 20 scale, traits of pronounced perfectionism with the scale adapted by Cox et al. from HF MPS, chronic fatigue syndrome as described after viral infections with the SOFA scale, functional disorders prior to infection with SARS-CoV-2, a former and/or current medical nomadism, a significant consumption of care. The quality of life is measured by the WHOQOL-BREF scale, anxious and/or depressive symptoms measured by the HAD scale, and sleep disorders assessed by the ISI scale .

ELIGIBILITY:
Inclusion Criteria:

* adults (18 years-old or older)
* having had a mild or moderate COVID-19 managed on an outpatient basis during the acute phase of the infection
* COVID-19 virologically confirmed or suspected on the basis of suggestive symptoms
* spontaneously consulting for post-COVID-19 symptoms and referred for neurological advice in our center
* with neurological clinical evaluation concluding that there is no differential diagnosis.

Exclusion Criteria:

* patients who were hospitalized during the acute phase of the infection
* suspected de novo neurological pathology unrelated to COVID-19
* patient refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients referred for neurology consultation to a referent neurologist in our center from may 2020 to may 2021
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
A positive diagnosis of SSD | 30 minutes
  all the following criteria: a PHQ15 score greater than or equal to 12 (criterion A); an SSD12 score greater than or equal to 23 (criterion B); an evolution of symptoms greater than or equal to four weeks for criterion C

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kachaner A, Lemogne C, Dave J, Ranque B, de Broucker T, Meppiel E. Somatic symptom disorder in patients with post-COVID-19 neurological symptoms: a preliminary report from the somatic study (Somatic Symptom Disorder Triggered by COVID-19). J Neurol Neurosurg Psychiatry. 2022 Aug 25:jnnp-2021-327899. doi: 10.1136/jnnp-2021-327899. Online ahead of print. PMID 36008115